CLINICAL TRIAL: NCT00527241
Title: Efficacy Trial of Raices Nuevas
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Joanne Klevens (U.S. Federal Agency)
Collaborators: University of Michigan (Other); The Community Health and Social Services Center, Inc. (Other)
Responsible Party: Sponsor-Investigator, Joanne Klevens, epidemiologist, Centers for Disease Control and Prevention
Organization: Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: U49CE000508 (NIH); IRB #4939
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Last update posted 2012-02-10 (Estimated); Status verified 2012-02

CONDITIONS: Intimate Partner Violence
Keywords: partner violence, spouse abuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: A (Experimental)
  Interventions: Behavioral: Raices nuevas
- 2 B (No Intervention): wait-listed for intervention to begin in 6 months

INTERVENTIONS:
Behavioral: Raices nuevas — 8 90-minute sessions (once a week) of problem-posing and facilitated discussion on respect, anger, support, trust, negotiating, partnership with your intimate partner.
  Arms: 1: A

SUMMARY:
This trial will test the impact of a culturally tailored and theory driven primary intimate partner violence prevention intervention with Spanish speaking Latino men.

DETAILED DESCRIPTION:
In this randomized controlled trial, Spanish speaking Latino men will be recruited from community church settings in Southwest Detroit and randomly assigned to: (a) an intimate partner violence prevention intervention or (b) a wait-list control condition. Latino men assigned to the intervention will receive, in a small group setting, an 8-session, primary intimate partner violence prevention intervention based on the Duluth model and culturally and linguistically tailored for Spanish speaking Latino men. Measures will be administered at pre-test, and at three and six months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Spanish speaking Latino men
* between the ages of 18 and 55
* in a stable relationship for at least the past three months

Exclusion Criteria:

* severely mentally impaired
* hearing impaired

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2006-11; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Perpetration of violence towards intimate partner | 3 and 6 months after completion of intervention

SECONDARY OUTCOMES:
intentions to abuse intimate partner | 3 and 6 months after completion of intervention
Beliefs, norms, and perceived self-efficacy | 3 and 6 months after completion of intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Community Health and Social Services Center (CHASS), Detroit, Michigan, United States